CLINICAL TRIAL: NCT00516165
Title: A Phase I/II Study of RAD001 in Advanced Hepatocellular Carcinoma
Brief Title: RAD001 in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-352
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; RAD001
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): Patients will receive RAD001 10 mg/day orally (6 weeks/cycle). Patients will be continued on treatment until disease progression, limiting toxicity, patient withdrawal of consent, or death.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Oral pills taken daily in a 42-day cycle (6 weeks). Cycles will be repeated every 42 days
  Other Names: Everolimus

SUMMARY:
Laboratory studies have shown that RAD001 can prevent cells from multiplying. Consequently, the study drug is being tested in medical conditions in which excessive cell multiplication (as in cancer) needs to be stopped. The main purpose of this research study is to find the highest dose of RAD001 that can be given safely (without causing severe side effects) and to learn the effects (good or bad) RAD001 has on participants with liver cancer.

DETAILED DESCRIPTION:
* Participants will be given a supply of the study drug RAD001 to be taken at home. They will be asked to take the study drug every morning on an empty stomach and will be given a study drug diary to record the time/date each time they take RAD001. Each 6 week period of time is called a cycle of study treatment.
* We are looking for the highest dose of RAD001 that can be given safely. Therefore not every participant will receive the same dose of RAD001.
* Participants will come to the clinic every other week. At each of these visits, a physical examination and blood tests will be performed.
* A CT and MRI will be repeated every 6 weeks during the first 3 cycles of treatment then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable of metastatic HCC. Patients must have prior core biopsy to confirm the diagnosis of HCC and have archived tissues available for correlative studies
* At least one measurable site of disease according to RECIST criteria that has not been previously irradiated. If it has had previous radiation to teh marker lesion(s), there must be evidence of progression since the radiation
* 0-2 prior systemic chemotherapy and biologic regimens for hepatocellular carcinoma
* Patients with prior chemoembolization history can participate in the study if the chemoembolization was performed more than 4 weeks ago and patients must have measurable disease outside of prior chemoembolization field
* 18 years of age or older
* Minimum of 4 weeks since any major surgery or completion of radiation
* Minimum of 4 weeks since completion of all prior systemic anticancer therapy
* ECOG performance status of 0-2
* CLIP score of equal to or less then 3
* Adequate bone marrow, liver and renal function as outlined in the protocol

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients with any severe and/or uncontrolled medical conditions or other condition that could affect participation in the study
* Known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Active, bleeding diathesis
* Women who are pregnant or breast feeding
* Patients who have received prior treatment with an mTor inhibitor
* Patients with known hypersensitivity to RAD001 or other rapamycins or its excipients
* History of non-compliance to medical regimens
* Patients with a positive dipstick for urine protein (reading of 2+ or greater) will then undergo a 24-hour urine collection for protein. If patients have a 2g or greater of protein/24hr, they will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 65 [33 to 81]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of RAD001 in Patients With Advanced Hepatocellular Carcinoma (HCC).
Time Frame: 2 years
Population: Patients with histologically confirmed measurable advanced Hepatocellular Carcinoma.
Measure: Number; unit: mg
Arm/Group | RAD001
Number analyzed (Participants) | 25
mg | 10
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p = 0.05, Kaplan Meier

2. Primary Outcome: Progression-free Survival Rate at 24 Weeks
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions"
  This information will be collected during two years of patient participation.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001
Number analyzed (Participants) | 28
months | 3.8 [2.1 to 4.6]
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p < 0.05, Kaplan-Meier

3. Secondary Outcome: Number of Patients With Adverse Events Who Were Treated With RAD001 for Advanced HCC
Description: Everolimus given at 10 mg/day as a single agent was well tolerated in patients with advanced HCC.
Time Frame: 2 years
Population: Patients with histologically confirmed measurable advanced HCC. The primary end points were determination of a safe dosage of everolimus and progression-free survival at 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001
Number analyzed (Participants) | 28
Participants | 28
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p < 0.05, Kaplan-Meier

4. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patient response
Arm/Group | RAD001
Number analyzed (Participants) | 28
percentage of patient response | 4 [0.9 to 19.6]
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p = 0.05, Kaplan-Meier

5. Secondary Outcome: Time to Progression
Description: 3.9 months with a CI of 21-
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | RAD001
Number analyzed (Participants) | 28
month | 3.9 [2.1 to 5.5]
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p = 0.05, Kaplan-Meier

6. Secondary Outcome: Overall Survival
Description: The median overall survival was 8.4 months (95% CI, 3.9-21.1 months). Only 2 ((8 %) patients were progression-free at 24 weeks. The study did not proceed to the second stage of the phase 2 portion of the study.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001
Number analyzed (Participants) | 28
months | 8.4 [3.9 to 21.1]
Statistical Analysis 1: Comparison: RAD001; Test type: Superiority or Other; p = 0.05, Kaplan-Meier

ADVERSE EVENTS:
Time Frame: October 2007 and June 2009; Participants were followed for this two year time period.
Description: 28 patients entered into the trial (9 in phase 1, 19 in phase 2) and all were evaluable for efficacy and toxicity based on intention-to-treat analysis. There were 18 men (64%) and 10 women (36%) with a median age of 65 years (range, 33-81 years).
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=28)
Grade 5-Death within 30 days. (General disorders) | 4 (4) — Unrelated
Grade 3 Encephalopathy-unrelated (Nervous system disorders) | 1 (1)
Grade 4 Anemia (Metabolism and nutrition disorders) | 1 (1) — Unlikely related
Grade 4 Thrombocytopenia (Metabolism and nutrition disorders) | 1 (1) — unrelated
Grade 4-Hypoxia (General disorders) | 1 — possibly related
Grade 4 Bilirubin (Gastrointestinal disorders) | 1 — unrelated
Grade 4 Hypophosphatemis (Blood and lymphatic system disorders) | 1 — unrelated
Respiratory failure (General disorders) | 1 — unrelated
Grade 4 elevated SGOT (Blood and lymphatic system disorders) | 1 — Unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=28)
Fatigue (General disorders) | 13 (52)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (48)
Anemia (Blood and lymphatic system disorders) | 11 (44)
Diarrhea (Gastrointestinal disorders) | 11 (44)
Leukopenia (Investigations) | 10 (40)
Platelets (Investigations) | 10 (40)
Aspartate transaminase (Investigations) | 9 (36)
Hyponatremia (Metabolism and nutrition disorders) | 9 (36)
Anorexia (Metabolism and nutrition disorders) | 9 (36)
Lymphopenia (Blood and lymphatic system disorders) | 8 (32)
Stomatitis (Gastrointestinal disorders) | 7 (28)
Rash (Skin and subcutaneous tissue disorders) | 7 (28)
Alanine transaminase (Investigations) | 6 (24)
Neutropenia (Investigations) | 5 (20)
Alkaline phosphatase (Investigations) | 4 (16)
Proteinuria (Investigations) | 4 (16)
Vomiting (Gastrointestinal disorders) | 4 (16)
Nausea (Gastrointestinal disorders) | 4 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (16)
Weight loss (Investigations) | 3 (12)
Acne rash (Skin and subcutaneous tissue disorders) | 3 (12)
Edema (Immune system disorders) | 3 (12)
Taste disturbance (Nervous system disorders) | 3 (12)
Hypoalbuminemia (Investigations) | 2 (8)
Hypokalemia (Investigations) | 2 (8)
Hypertriglyceridemia (Investigations) | 2 (8)
Fever without neuropenia (Investigations) | 2 (8)
Constipation (Gastrointestinal disorders) | 2 (8)
Nose bleeds (Investigations) | 2 (8)
Cough (General disorders) | 2 (8)
Insomnia (General disorders) | 2 (8)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (8)
Pain (Gastrointestinal disorders) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No